CLINICAL TRIAL: NCT00423553
Title: Modifying Tolerance to Ischemic Injury in Human Atrial Tissue
Brief Title: Collection of Heart Tissue Sample During Open Heart Surgery
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070057; 07-H-0057
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Ischemia
Keywords: Nitrite and Cytoprotection; Ischemic Preconditioning; Atrial Trabeculae Contractile Function; Ischemia
MeSH Terms: conditions — Ischemia

SUMMARY:
This study will collect heart tissue that is routinely removed and discarded during open-heart surgery. The Cardiology Branch of the NHLBI is conducting a variety of laboratory experiments that require a sample of heart tissue. A segment of tissue is routinely cut out of the right atrial appendage of the heart during open-heart surgery to allow the heart-lung bypass machine to be attached to the heart for protection during surgery. This small tissue sample is not re-attached after the bypass machine is removed, but usually destroyed as medical waste.'

People between 18 and 80 years of age who are scheduled to undergo coronary artery bypass surgery or aortic valve replacement surgery may be eligible for this study.

Participants donate the right atrial appendage of the heart, which would normally be destroyed after their open-heart surgery. The tissue will be used by NHLBI investigators in studies directed at learning how to make the heart less sensitive to damage from a heart attack. The samples may be used, for example, to evaluate the effectiveness of known therapies, refine treatment approaches, identify potential new therapies, or explore opportunities for disease prevention.

DETAILED DESCRIPTION:
Transient non-lethal ischemia followed by reperfusion activates a cell survival program resulting in increased tolerance to subsequent ischemic injury. This biological phenomenon is termed ischemic preconditioning and is a powerful cell survival program that is operational in the human heart. This program is triggered by signaling intermediates activated in response to the transient ischemia/hypoxia and reperfusion of preconditioning. Characterization of these signaling intermediates should enable us to identify therapeutic agents to augment tissue tolerance to ischemia.

Interestingly, nitrite, which is an endogenous reservoir for nitric oxide (NO), undergoes bioconversion to NO via hypoxia-dependent signaling. Whether nitrite accumulation and bioconversion are components of the ischemic preconditioning program is unknown. Recently Dr. Gladwin and colleagues in the Vascular Medicine Branch unequivocally demonstrated that exogenous nitrite administration is cytoprotective against ischemia-reperfusion injury in murine liver and heart and in the canine heart. Establishing a mechanistic link between the ischemic preconditioning program and nitrite biology would promote nitrite as an attractive compound for future therapeutic interventions. To evaluate this link, we propose to use cardiac right atrial appendage tissue that is routinely excised to facilitate right atrial cannulation for heart-lung bypass. This excised tissue is then usually discarded as medical waste.

We hypothesize that nitrite administration to atrial tissue in an ex-vivo study will demonstrate increased tolerance to ischemic stress compared to atrial tissue not exposed to nitrite. Furthermore, we propose that this cytoprotective effect of nitrite administration will demonstrate equivalency to cytoprotection in response to ischemic preconditioning. Finally, we would employ this tissue to identify nitrite mediated genomic, proteomic and metabolomic modifications in human myocardium, thereby identifying the biological programs orchestrating the cytoprotective properties of nitrite in the human heart.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must be 18-80 years of age.

Subjects must provide informed, written consent to donate tissue that would otherwise be discarded post-cardiac surgery.

Subjects undergoing elective coronary artery bypass surgery and or aortic valve replacement surgery.

EXCLUSION CRITERIA:

Subjects currently on oral sulfonylurea therapy for diabetes mellitus

Subjects in atrial fibrillation or having had a history of atrial fibrillation in the 2-week period prior to surgery

Subjects in clinical right heart failure as evidenced by greater than trace pedal edema, an elevated JVP and or by evidence of hepatic congestion.

Subjects unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 2007-01-11; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (1):
- Suburban Hospital, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gladwin MT, Shelhamer JH, Schechter AN, Pease-Fye ME, Waclawiw MA, Panza JA, Ognibene FP, Cannon RO 3rd. Role of circulating nitrite and S-nitrosohemoglobin in the regulation of regional blood flow in humans. Proc Natl Acad Sci U S A. 2000 Oct 10;97(21):11482-7. doi: 10.1073/pnas.97.21.11482. PMID 11027349